CLINICAL TRIAL: NCT04858269
Title: Phase II Study of First Line Weekly Chemo/Immunotherapy for Metastatic Head/Neck Squamous Cell Carcinoma Patients
Brief Title: First Line Weekly Chemo/Immunotherapy for Metastatic Head/Neck Squamous Cell Carcinoma Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00072117; WFBCCC 60121 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Head Neck Cancer; Metastatic Squamous Cell Carcinoma; Oral Cavity Squamous Cell Carcinoma; Oropharynx Squamous Cell Carcinoma; Hypopharynx Squamous Cell Carcinoma; Larynx Squamous Cell Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination of Chemotherapy and Immunotherapy (Experimental): The intervention will be administered on an outpatient basis. The treatment regimen will consist of combination chemotherapy and immunotherapy administered as: Pembrolizumab PLUS Carboplatin PLUS Paclitaxel.
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg intravenously (IV) on day 1 of each 3-week cycle
Drug: Carboplatin — Carboplatin dosed for area under the curve (AUC) 1.5 IV on days 1, 8, 15 of each 3-week cycle
Drug: Paclitaxel — Paclitaxel 45 mg/m2 on days 1, 8, 15 of 3-week cycle.

SUMMARY:
The purpose of this research is to see what effects the treatment regimen chemotherapy (carboplatin and paclitaxel) plus immunotherapy (pembrolizumab), has on patients who have been diagnosed with head/neck squamous cell carcinoma and are unable to take the drug 5-fluorouracil

DETAILED DESCRIPTION:
Primary Objective: To determine if six (6) cycles of pembrolizumab with weekly carboplatin and paclitaxel for the 1st line treatment of metastatic head/neck squamous cell carcinoma patients increases the radiographic response rate as compared to the historical rate for pembrolizumab alone.

Secondary Objective(s):

* To determine if six (6) cycles of pembrolizumab with weekly carboplatin and paclitaxel for the 1st line treatment of metastatic head/neck squamous cell carcinoma patients increases median overall survival (OS) as compared to the historical rate reported for pembrolizumab alone.
* To determine if six (6) cycles of pembrolizumab with weekly carboplatin and paclitaxel followed by pembrolizumab alone for the 1st line treatment of metastatic head/neck squamous cell carcinoma patients increases the median progression-free survival (PFS) as compared to the historical rate reported for pembrolizumab alone.
* To determine the toxicity profile of six (6) cycles of pembrolizumab with weekly carboplatin/paclitaxel/pembrolizumab alone for the 1st line treatment of metastatic head/neck squamous cell carcinoma patients, measured as the proportion of patients with discontinuation of any study drug due to any adverse event of any cause, as compared to the historical proportion reported for platinum/5FU/ pembrolizumab (33%).

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 and carboplatin IV and paclitaxel IV on days 1, 8, and 15. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 21 days and then every 28 days for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or metastatic squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, larynx or neck node with occult primary but suspected to be non-cutaneous head/neck that is incurable by local therapies (i.e. radiation or surgery) and either locoregionally advanced or with at least one distant metastasis.
* Histologic or cytologic confirmation of malignancy by pathology report.
* Not a candidate for infusional 5FU (mucositis, 5-day infusional pump not feasible, patient refusal, other).
* 18 years old or greater.
* ECOG performance status of 0-2.
* Life expectancy of greater than 3 months.
* Patients must have normal organ and marrow function as defined: Absolute neutrophil count greater than or equal to 1,000/mcL, platelets greater than or equal to 75,000/mcL, total bilirubin less than or equal to 2 mg/dL
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).

Exclusion Criteria:

* No prior systemic cancer-directed therapy administered in the recurrent or metastatic setting. Prior treatments are allowed if they were administered with curative intent prior to incurable progression of disease. Prior treatments for other cancers are also allowed.
* Untreated, symptomatic central nervous system (CNS) metastases.
* Active autoimmune disease requiring systemic immunosuppression.
* History of autoimmune pneumonitis requiring high-dose systemic steroids (equivalent prednisone >20 mg/day for >1 week).
* History of greater than or equal to Grade 3 hypersensitivity reaction to carboplatin or paclitaxel.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because paclitaxel and carboplatin are Class D agents with significant potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these drugs, breastfeeding should be discontinued during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Response Rate | At 18 weeks on study
  Using RECIST 1.1 will be defined as the percentage of analyzed participants with a complete response - defined as disappearance of all target lesions; or partial response - defined as decrease by ≥ 30% in sum of longest diameter of target lesions when compared to the historical objective response rate (19%) reported for pembrolizumab alone; stable disease (SD): Not meeting criteria for CR, PR, or PD; progressive disease (PD): Increase by ≥ 20% in sum of longest diameter of target lesions or the appearance of one or more new lesions.

SECONDARY OUTCOMES:
Overall Survival | Up to 2 years
  Median survival rate will be defined as the time from study registration to death due to any cause and as compared to the historical median reported for pembrolizumab alone. The Kaplan-Meier method will be used to generate survival curves with the intention-to-treat population. Data for patients who are alive or lost to follow-up will be censored for overall survival at the date they were last known to be alive
Progression-Free Survival | Up to 2 years
  Median progression-free survival (PFS) defined as the time from study registration to the first documented progressive disease (PD) per RECIST v1.1 criteria (defined as increase by ≥ 20% in sum of longest diameter of target lesions or the appearance of one or more new lesions) based on non-blinded central imaging or else death due to any cause, whichever occurred first; and as compared to the historical value reported for pembrolizumab alone. The Kaplan-Meier method will be used to generate survival curves with the intention-to-treat population.
Number of Participants with Discontinuation of Study Drug due to Adverse Effects of Any Cause | Up to 18 weeks
  Participants with discontinuation of any study drug due to adverse events of any cause before 18 weeks as compared to the historical value reported for platinum/5FU/pembrolizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lycan, DO, Principal Investigator — Wake Forest Baptist Health Sciences
Locations (1):
- Wake Forest Baptist Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No